CLINICAL TRIAL: NCT03392363
Title: Diagnosing Respiratory Disease in Children Using Smartphone Recordings of Cough Sounds 2
Brief Title: Diagnosing Respiratory Disease in Children Using Cough Sounds 2
Acronym: SMARTCOUGH-C-2
Status: Completed | Type: Observational
Sponsor: ResApp Health Limited (Industry)
Collaborators: Massachusetts General Hospital (Other); The Cleveland Clinic (Other); Baylor College of Medicine (Other); Baim Institute for Clinical Research (Other)
Responsible Party: Sponsor
Other Study IDs: 17001
Record Dates: First submitted 2017-12-29; First posted 2018-01-05 (Actual); Last update posted 2018-11-08 (Actual); Status verified 2018-11

CONDITIONS: Pneumonia; Bronchiolitis; Asthma Exacerbation; Croup; Reactive Airway Disease; Upper Respiratory Disease; Viral Lower Respiratory Tract Infections; Lower Respiratory Disease
MeSH Terms: conditions — Pneumonia; Bronchiolitis; Croup; Pulmonary Disease, Chronic Obstructive; Respiration Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Device: Recordings of Infants and Children's Cough Sounds — Smartphone recordings of the cough sounds of infants and children presenting to a participating site with signs or symptoms of respiratory disease.

SUMMARY:
The purpose of this prospective study is to evaluate the efficacy of the ResAppDx software application in the diagnosis of childhood acute respiratory disease, including pneumonia, bronchiolitis, asthma/reactive airways disease, croup, lower respiratory tract disease (LRTD), viral lower respiratory tract infection (vLRTI), and upper respiratory tract disease (URTD).

ELIGIBILITY:
Inclusion Criteria:

* Infant or child aged greater than 29 days up to and including their 12th birthday (infant and children pediatric subgroups as defined in Guidance for Industry and Food and Drug Administration Staff: Premarket Assessment of Pediatric Medical Devices dated March 24, 2014)
* Presenting to the study site (an outpatient facility, an urgent care center, an Emergency Department, or inpatient ward within 24 hours of admission) with current signs or symptoms of respiratory disease including cough, wheezing, stridor, chest in-drawing/retractions, difficulty breathing, fast breathing, nasal congestion/rhinorrhea, abnormal lung sounds on exam or cyanosis/hypoxemia.
* Onset of symptoms within past 14 days
* Outpatient or inpatient within 24 hours of admission
* Coughing spontaneously or able to cough voluntarily

Exclusion Criteria:

* Lack of a signed consent form from parent or legal guardian
* Lack of signed assent form for children aged 7 years or older who, in the opinion of the investigator, is able to provide assent based on their age, maturity or psychological state.
* Need for mechanical ventilatory support ((including invasive, CPAP, or BiPAP)) or high flow nasal cannula
* History of structural airways abnormalities, tracheobronchomalacia, or vocal cord abnormalities (e.g. laryngomalacia, tracheomalacia, or bronchomalacia)
* Any medical contraindication to voluntary cough, including the following (only enroll if coughing spontaneously): severe respiratory distress, history of pneumothorax, eye/chest/abdominal surgery in past 3 months, hemoptysis in the past month
* Too medically unstable to participate in study per treating clinician
* Subject previously enrolled in SMARTCOUGH-C-2 study
* Tracheostomy present or tube placed

Ages: 29 Days to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients with signs or symptoms of respiratory disease presenting to participating Emergency Departments, Urgent Care Clinics, Outpatient Clinics or an Inpatient Ward within 24 hours of admission.
Sampling Method: Non-Probability Sample
Enrollment: 1470 (Actual)
Dates: Start 2018-01-05 (Actual); Primary Completion 2018-10-19 (Actual); Study Completion 2018-10-19 (Actual)

PRIMARY OUTCOMES:
Diagnosis of pneumonia | 6 months
  Positive percent agreement and negative percent agreement to diagnose and rule out pneumonia as compared with (1) World Health Organization (WHO) Primary Endpoint Pneumonia (PEP) plus clinical pneumonia, (2) WHO PEP or Other Infiltrate plus clinical pneumonia, (3) Clinical pneumonia alone
Diagnosis of other childhood respiratory diseases | 6 months
  Positive percent agreement and negative percent agreement to diagnose and rule out: lower respiratory tract disease (i.e. respiratory condition occurring below the level of the larynx), viral lower respiratory tract infection, bronchiolitis, asthma/reactive airways disease, upper respiratory tract disease, and croup.

CONTACTS AND LOCATIONS:
Overall Officials: Peter P Moschovis, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Cleveland Clinic Children's, Cleveland, Ohio
  - Texas Children's Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: No